CLINICAL TRIAL: NCT05965843
Title: Research on the Intervention, Prognosis and Mechanism of Novel Coronavirus Infection in Patients With Underlying Diseases
Brief Title: Intervention, Prognosis and Mechanism of Covid-19 Infection in Patients With Underlying Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023IITXG01
Record Dates: First submitted 2023-07-27; First posted 2023-07-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Chronic Liver Disease; Malignant Tumor; Autoimmune Diseases; Healthy
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- chronic liver disease: No additional interventions for this group.
  Interventions: Other: underling disease
- malignant tumor: No additional interventions for this group.
  Interventions: Other: underling disease
- autoimmune disease: No additional interventions for this group.
  Interventions: Other: underling disease
- medical staff: No additional interventions for this group.
  Interventions: Other: underling disease

INTERVENTIONS:
Other: underling disease — Nowadays Covid-19 virus has become milder than before however severe outcomes still happen in people with underlying diseases after infection.
  For example, previous research indicated cirrhosis was an independent predictor for COVID-19 mortality.
  More efforts shoud be make to explore the association between underlying diseases and severe COVID-19.

SUMMARY:
The goal of this observational study is to explore the influence of Covid-19 infection and risk factors of severe outcomes in vulnerable population including patients with chronic liver disease, malignant tumor, autoimmune disease, medical staff.

The main questions it aims to answer are:

1. The clinical characteristics of vulnerable population after Covid-19 infection.
2. Risk factors for severe illness in vulnerable groups after infection with the Covid-19.
3. The impact of Covid-19 infection on the progression of underlying diseases.

Information of participants will be collected such as gender, age, underlying diseases, medication status, vaccination status, clinical and biochemical indicators.

Researchers will compare the mild and severe outcomes after Covid-19 infection to identify the "truly vulnerable" population and explore the potential mechanism and intervention for these population.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before enrollment, and be able to complete the research according to the requirements of the research protocol.
2. Enrolled patients need to have basic diseases, including chronic liver disease, chronic kidney disease, chronic lung disease, solid tumors, AIDS, rheumatic immune diseases, diabetes, etc.
3. When entering the group, patients with new crowns need to be confirmed by evidence of a positive test for new coronavirus nucleic acid (CT value <35) or a positive test for new coronavirus antigen.

Exclusion Criteria:

1. Participate in clinical trials of other investigational drugs or medical devices within 3 months before screening, and take experimental drugs or use medical devices.
2. Positive pregnancy test during lactation or screening period.
3. Subjects who, in the investigator's opinion, have other factors that are not suitable for participating in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population was population with underling disease from single-centre and medical staff from multiple centers in Chongqing.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality in patients with underline disease after Covid-19 infection. | 30 days
  All-cause mortality is a measure of the total number of deaths from any cause.

SECONDARY OUTCOMES:
Severe disease in patients with underline disease after Covid-19 infection. | 48weeks
  Severe disease include severe Covid-19 and/or progression of underlying disease.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Hu, PhD., Study Director — The Second Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: Undecided